CLINICAL TRIAL: NCT01816711
Title: Vitamin D Levels in Frail Elderly Patients With a Hip Fracture
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: HFVD2012; 2007-58-0010 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2013-04

CONDITIONS: Hip Fracture; Vitamin D Deficiency
Keywords: Frail elderly; Hip fracture; Vitamin D; Geriatrics
MeSH Terms: conditions — Hip Fractures; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hip fracture, Frail elderly, Non-supplemented: Frail elderly with a hip fracture who did not received vitamin D supplementation
- Hip fracture, Frail elderly, Supplemented: Frail elderly with a hip fracture who received vitamin D supplementation

SUMMARY:
The purpose of this study is to assess whether all frail elderly admitted with hip fracture has a vitamin D deficiency, and if s-25(OH)D deficiency increases the risk of hip fracture in frail elderly.

Frail elderly are defined as being 65 years of age or older, and living in nursing homes or senior housings.

The investigators' hypotheses state that:

1. Frail elderly with hip fractures will have a suboptimal level of vitamin D.
2. Frail elderly with hip fractures are more likely to have a suboptimal level of vitamin D than frail elderly without any hip fractures during the last ten years.

DETAILED DESCRIPTION:
The study examined frail elderly patients, defined as 65 of age or older and living nursing homes or senior housings.

Cases where taken from a Randomised Controlled Trial (NCT01102010), where the included where frail elderly admitted with a hip fractures to the Orthopaedic Surgery Ward at Aarhus University Hospital.

Controls were frail elderly, without a hip fracture in the previous ten years, admitted to the Geriatric Ward at Aarhus University Hospital.

The investigators will look at all eligible patients' files and record their serum-25(OH)D levels upon admission.

According to sample size calculations 92 patients are needed in the case group, and 138 patients in the control group.

The inclusion period will be from the 18th of January 2010 to the 1st of October 2012 for both groups.

ELIGIBILITY:
Inclusion Criteria, Cases:

* Aged 65 or older
* Living in nursing home or senior housing
* Admitted with hip fracture to the Orthopaedic Ward, Aarhus University Hospital

Exclusion Criteria, Cases:

* No serum-25(OH)D measurement upon admission

Inclusion Criteria, Controls:

* Aged 65 or older
* Living in nursing home or senior housing
* Admitted to the Geriatric Ward, Aarhus University Hospital

Exclusion Criteria, Controls:

* No serum-25(OH)D measurement upon admission
* Hip fracture in the previous ten years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cases were frail elderly admitted with a hip fracture to the Orthopaedic Ward at Aarhus University Hospital in the period: 18th of January 2010 to the 1st of October 2012.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Reasearch Unit, Geriatric Department, Aarhus University Hospital, Aarhus, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Hip Fracture, Frail Elderly, Non-supplemented: Cases: Frail elderly with a hip fracture who did not receive vitamin D supplementation
Period: Overall Study
Arm/Group | Hip Fracture, Frail Elderly, Non-supplemented | Hip Fracture, Frail Elderly, Supplemented
Started | 121 | 83
Completed | 121 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hip Fracture, Frail Elderly, Non-supplemented: Frail elderly with a hip fracture who did not receive vitamin D supplementation
- Total: Total of all reporting groups
Arm/Group | Hip Fracture, Frail Elderly, Non-supplemented | Hip Fracture, Frail Elderly, Supplemented | Total
Number analyzed (Participants) | 121 | 83 | 204
Age, Continuous [Mean (Full Range); unit: years] | 87 [71 to 100] | 83 [65 to 98] | 87 [65 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 62 | 150
  Male | 33 | 21 | 54
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 121 | 83 | 204
Senior housing [Count of Participants; unit: Participants] | 44 | 38 | 82
Nursing home [Count of Participants; unit: Participants] | 77 | 45 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suboptimal and Optimal Levels of Vitamin D (Serum-25(OH)D)
Description: Serum-25(OH)D was measured in a blood sample as an indicator of Vitamin D status
Time Frame: Upon admission
Measure: Count of Participants; unit: Participants
Arm/Group | Hip Fracture, Frail Elderly, Non-supplemented | Hip Fracture, Frail Elderly, Supplemented
Number analyzed (Participants) | 121 | 83
Participants
  Suboptimal level (<75nmol/l) | 106 | 42
  Optimal level (>75nmol/l) | 15 | 41

ADVERSE EVENTS:
Arm/Group | Hip Fracture, Frail Elderly, Non-supplemented | Hip Fracture, Frail Elderly, Supplemented
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/83
Other Adverse Events (participants affected / at risk) | 0/121 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes